CLINICAL TRIAL: NCT06747598
Title: Efficacy Evaluation of Using Finger Stick Peripheral Blood for Point of Care Pregnancy Testing
Acronym: POCPREG
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0755-24-EP
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy Testing
Keywords: POC pregnacy testing serum
MeSH Terms: interventions — Pregnancy Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- POC serum pregnancy test arm: Enrolled participants will provide a peripheral serum specimen for POC pregnancy testing
  Interventions: Diagnostic Test: pregnancy test

INTERVENTIONS:
Diagnostic Test: pregnancy test — POC pregnancy testing using peripheral serum

SUMMARY:
To evaluate the efficacy of using peripheral blood for POC pregnancy testing in known pregnant participants.

DETAILED DESCRIPTION:
Point of care (POC) pregnancy tests are designed for use with a urine specimen. However, the timely collection of a urine specimen is solely dependent on the patient's need to urinate which can delay the initiation of subsequent care activities. Furthermore, when considering the limitations of urine POC testing in wilderness scenarios, collecting a urine specimen from an injured person may not be a viable option. The literature has demonstrated blood as a viable alternative specimen for use with POC pregnancy testing with a sensitivity of 95.8%. Based on a literature review, these studies used blood specimen that were pre-collected into a serum collection vial. The study postulates the use of peripheral blood via a finger stick has multiple benefits such as 1) eliminating the need to wait for urine, 2) expedite the serum collection process as compared to a venipucture, 3) allow for testing in non-traditional scenarios such as wilderness medicine or mass casualty/gathering scenarios, and 4) minimizing the amount of blood required as compared to a traditional 3-5 ml serum collection vial. Data from this pilot study will provide valuable insight on the potential use of this testing method to inform future studies and treatment protocols for the above mentioned scenarios.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant female, 19 years or older, being seen at the Nebraska Medicine OB/GYN clinic

Exclusion Criteria:

* Does not meet inclusion criteria

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant Female
Study Population: 30 confirmed pregnant patients who present for their routine care visit to confirm efficacy of finger stick pregnancy test
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
POC serum pregnancy testing | One time test at time of enrollment
  A peripheral serum specimen will be used to test for pregnancy using a POC test. Outcome will be positive or negative

CONTACTS AND LOCATIONS:
Overall Officials: Thanh T Nguyen, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-08-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT06747598/ICF_000.pdf